CLINICAL TRIAL: NCT02400866
Title: A Randomized Study of Olanzapine for the Prevention of CINV in Patients Receiving Moderately Emetogenic Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korean South West Oncology Group (Network)
Responsible Party: Principal Investigator, Hwan Jung Yun, Professor, Korean South West Oncology Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSWOG 15-01
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Cancer
Keywords: cancer patients receiving moderately emetogenic chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): palonosetron + dexamethasone + placebo
- Experimental (Experimental): palonosetron + dexamethasone + olanzapine
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine
  Arms: Experimental

SUMMARY:
This aim of study is to evaluate the safety and efficacy of olanzapine for the prevention of chemotherapy-induced nausea and vomiting in patients receiving moderately emetogenic chemotherapy by a randomized, double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* over 19 years of age
* no history of receiving moderately or highly emetogenic chemotherapy during last 6 months, and is to receive a first course of MEC including one or more of following agents: Carboplatin, Cyclophosphamide ≤ 1,500 mg/m2, Daunorubicin, Doxorubicin < 60 mg/m2, Epirubicin ≤ 90 mg/m2, Irinotecan, Oxaliplatin, Melphalan, Methotrexate ≥ 250 mg/m2
* ECOG performance status 0-2
* predicted life expectancy ≥ 3 months
* adequate bone marrow, kidney, and liver functionas evidenced by: ANC ≥ 1,500/mm3, platelet count ≥ 100,000/mm3, total bilirubine ≤ 2 x ULN, AST ≤ 3 x ULN, ALT ≤ 3 x ULN (for subjects with known liver metastases, total bilirubin ≤ 3 x ULN, AST ≤ 5 x ULN, ALT ≤ 5 x ULN), Creatinine ≤ 1.5 x ULN or Ccr ≥ 50 ml/min
* no episodes of nausea and vomiting during last 24 hours before enrollment
* subjects provides written informed consent

Exclusion criteria:

* subjects with uncontrolled neuro-psychiatric disease (alcohol abuse, seizure, psychosis etc) except malignant tumor
* subject is scheduled to receive highly emetogenic chemotherapeutic agents: Doxorubicin or Epirubicin + cyclophosphamide, Cisplatin ≥ 50 mg/m2, Carmustine > 250 mg/m2, Cisplatin ≥ 50 mg/m2, Cyclophosphamide > 1,500 mg/m2, Dacarbazine, Doxurubicine ≥ 60 mg/m2, Epirubicine > 90 mg/m2, Ifosfamide ≥ 2 g/m2 per dose, Mechlorethamine, Streptozocin
* contraindication to the administration of palonosetron, dexamethasone, and olanzapine due to hypersensitivity or any other reasons
* subject has severe cognitive impairment
* subjects has symptomatic or uncontrolled brain metastasis or brain tumor
* female subjects of childbearing potential who dose not agree to use a proper contraceptive methods or to limit breast feeding
* subject has taken the following agents: risperidone, quetiapine, clozapine, phenothiazine, butyrophenone, 5-HT3 antagonist, bezamides, domperidone, cannabinoids, NK1 antagonist, bezodiazepines
* subject has a plan to receive other chemotherapy, abdomial radiation, surgery, or immunotherapy
* any history of arrhythmia, uncontrolled congestive heart failure, acute myocardial infarction durting last 6 months
* history of uncontrolled diabetes
* subject who has used any investigational drugs within 30 days of randomization

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-11 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
complete response rate for the acute phase (0-24 hours) after chemotherapy | during 24 hours after first cycle of moderately emetogenic chemotherapy (MEC)

SECONDARY OUTCOMES:
complete response rate for the delayed phase (24-120 hours) and overall phase (0-120 hours) after chemotherapy | during 0-120 hours after first cycle of MEC
no vomiting for the overall phase | during 0-120 hours after first cycle of MEC
significant emesis for the overall phase | during 0-120 hours after first cycle of MEC
numbers and time for rescue medicaions | during 0-120 hours after first cycle of MEC
effects on quality of life by FLIE questionnaire | during 0-120 hours after first cycle of MEC